CLINICAL TRIAL: NCT03401593
Title: Long Term Evaluation and Management of Atrial Fibrillation in Pacemaker Patients (AF-pacemaker Tx Study)
Brief Title: Long Term Evaluation and Management of Atrial Fibrillation in Pacemaker Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-1028
Record Dates: First submitted 2017-12-27; First posted 2018-01-17 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Permanent Pacemaker Implantation
Keywords: ablation; atrial fibrillation; stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ablation (Active Comparator): Patients in this group are treated with radio-frequency catheter ablation.
  Interventions: Drug: midazolam with fentanyl
- non-ablation (No Intervention): Patients in this group are treated with rate control medications (e.g., beta blocker, calcium channel blocker, and digitalis) and anti-arrhythmic drugs. They also can be treated with DC cardio-version.

INTERVENTIONS:
Drug: midazolam with fentanyl — Radio-frequency catheter ablation is performed in the post-absorptive state after sedation with midazolam and fentanyl. Multipolar catheters were positioned in the coronary sinus, His, and the right atrium. The three-dimensional LA geometry was reconstructed using a CARTO or NavX electroanatomical mapping system. Circumferential pulmonary vein isolation was performed in all patients using a irrigated-tip catheter. A circular mapping catheter was used to confirm the isolation of the pulmonary veins. Successful ablation was defined by the elimination of all the pulmonary vein potentials along the antrum or inside the veins. If the AF was not terminated after elimination of all the pulmonary vein potentials, linear ablation and complex fragmented atrial electrogram ablation were performed.
  Arms: ablation

SUMMARY:
This study is prospective randomized study which was performed in multicenter (General Hospital) in Korea. Inclusion criteria is patients who developed atrial fibrillation/flutter/tachycardia after pacemaker implantation among AF-pacemaker study (ClinicalTrials.gov Identifier: NCT03303872). The purpose is to investigate the recurrence rate of AF/AFL/AT in both groups after randomization for 60 months (5 years) in patients post pacemaker implantation and assess long term clinical results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who developed atrial fibrillation/flutter/tachycardia after pacemaker implantation among AF-pacemaker study (ClinicalTrials.gov Identifier: NCT03303872).
* Age: 18-80 years
* Patients eligible for the indications for permanent pacemaker implantation in accordance with 2016 revised Korean indication guideline on cardiac pacemaker implantation
* Estimated percentage of atrial pacing >40% under sinus rhythm (LR≥60bpm, close hysteresis and rest rate)
* Estimated percentage of ventricular pacing >40% under sinus rhythm (LR≥40bpm, DDD pacing, close hysteresis and rest rate)
* Patients who are willing to sign the informed consent.
* Patients who are willing to receive the implantation and post-operative follow-up.

Exclusion Criteria:

* Persistent or permanent AF
* Severe hepatic and renal insufficiency (AST or ALT ≥ three times of normal upper limit; SCr > 3.5 mg/dl or Ccr < 30ml/min)
* Thyroid gland dysfunction
* Pregnancy
* Malignant tumor
* Severe organic heart disease (such as moderate to severe mitral regurgitation, severe valvular regurgitation and stenosis, dilated cardiomyopathy, hypertrophic cardiomyopathy, severe heart valve disease)
* Life expectancy < 12 months
* Patients unable or unwilling to cooperate in the study procedures.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of AF/AFL/AT in both groups | 1 year after randomization
  recurrence of AF/AFL/AT evaluated using device interrogation
Recurrence rate of AF/AFL/AT in both groups | 6-month follow up to 5 years
  recurrence of AF/AFL/AT evaluated using device interrogation

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 1 year after randomization
  cardiac function evaluated using echocardiography
Left atrial diameter | 1 year after randomization
  cardiac function evaluated using echocardiography
Stroke | at least 1 year after randomization
  ischemic and hemorrhagic stroke
Stroke | 6-month follow up to 5 years
  ischemic and hemorrhagic stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea